CLINICAL TRIAL: NCT00461929
Title: Are the Secondary Chromosome Abnormalities Seen in Chronic Myeloid Leukemia (CML) Cells Induced to Ph-Chromosome Negativity by Imatinib a Result of Chromosome Instability or a Side Effect of the Therapy - a Study in GIST (Gastrointestinal Stromal Cell Tumors) Patients Treated With Imatinib.
Brief Title: Chromosome Abnormalities in Chronic Myeloid Leukemia (CML) on Imatinib. GIST Patients on Imatinib
Acronym: GIST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study terminated 12Feb09 due to low recruitment
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Mount Sinai Hospital, Canada (Other); Novartis (Industry)
Responsible Party: Dr. Jeff Lipton, University Health Network, Princess Margaret Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CST1571ACA10 GIST
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Myeloid Leukemia; Gastrointestinal Stromal Cell Tumors; Chromosome Abnormality
Keywords: chronic myeloid leukemia; gastrointestinal stromal cell tumors; chromosome abnormality; imatinib; bone marrow aspiration
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Chromosome Aberrations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bone marrow aspiration

SUMMARY:
In order to distinguish between clonal instability driven by imatinib in CML and actual changes with secondary clones induced by imatinib we would like to investigate the karyotype of non-CML patients treated with imatinib such as GIST patients.

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is a myeloproliferative disorder characterized by the presence of the Philadelphia (Ph) chromosome - a t(9:22) translocation that results in the production of a BCR/ABL fusion protein with Abl kinase activity.

Imatinib mesylate (Gleevec) specifically targets a limited set of protein tyrosine kinases - ABL, Arg (Abl-related gene), c-Kit, platelet-derived growth factor receptor (PDGF-R) - and their oncogenic forms, most notably BCR/ABL Imatinib is also a potent inhibitor of a receptor-type c-Kit tyrosine kinase. Therefore imatinib was examined for therapeutic efficacy against malignant gastro-intestinal stromal tumors (GIST) Recent articles have drawn attention to the development of new Ph-negative, cytogenetically unrelated clones after therapy of Ph-positive CML with imatinib. Trisomy 8 and monosomy 7 are the most frequent defects, but other aberrations have also been reported. Some of these cytogenetic abnormalities are associated with acute myeloid leukemia and MDS.

ELIGIBILITY:
Inclusion Criteria:

* GIST patient on Imatinib for more than 12 months

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
~ presence or absence of genetic abnormality as seen in CML patients on imatinib

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Lipton, MD, Principal Investigator — University Health Network, DMOH; Martin Blackstein, MD, Study Director — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario